CLINICAL TRIAL: NCT01627067
Title: Circulating FGF21 Levels and Efficacy of Exemestane, Everolimus and Metformin in Postmenopausal Women With Hormone Receptor Positive Metastatic Breast Cancer and BMI >/= 25
Brief Title: Exemestane-RAD001-Metformin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Komen Foundation Funding Terminated
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1239; NCI-2012-01164 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hormone Receptor Positive Metastatic Breast Cancer; Hormone-sensitive; Postmenopausal; Body Mass Index; BMI; Everolimus; Afinitor; RAD001; Exemestane; Aromasin; Metformin
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; exemestane; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Everolimus + Exemestane + Metformin (Experimental): Patients take one 25 mg tablet of exemestane once daily, everolimus 10 mg orally per day and metformin 500 mg orally per day for three days. If there are no dose limiting toxicities, dose of metformin will be increased by 500 mg orally every three days to reach the target dose of 1,000 mg orally twice daily. Drugs will be taken immediately after a meal at the same time each day.
  Interventions: Drug: Everolimus; Drug: Exemestane; Drug: Metformin

INTERVENTIONS:
Drug: Everolimus — 10 mg by mouth once daily.
  Other Names: Afinitor; RAD001
Drug: Exemestane — 25 mg by mouth once daily.
  Other Names: Aromasin
Drug: Metformin — 500 mg by mouth per day for three days. If there are no dose limiting toxicities, the dose of metformin will be increased by 500 mg orally every three days to reach the target dose of 1,000 mg orally twice daily.

SUMMARY:
The goal of this clinical research study is to learn if exemestane and everolimus combined with metformin can help to control breast cancer in patients who are obese or overweight and post-menopausal with hormone-receptor-positive breast cancer that has spread to other parts of the body.

Exemestane is designed to decrease the ability of estrogen to help cancer cells grow. This could cause the cancer cells to die.

Metformin is commonly used to control blood sugar levels in patients with diabetes. It is designed to lower insulin levels, which may slow or stop the growth of breast cancer cells.

Everolimus is designed to block cells from dividing. This may cause cancer cells to die. Everolimus may also stop the growth of new blood vessels that help tumors grow.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take an exemestane and everolimus tablet by mouth every day. You will also take tablets of metformin by mouth 2 times a day. The drugs should be taken at about the same time each day.

The study drugs will be given in 28-day cycles.

Study Visits:

On Day 1:

* You will have a physical exam, including a measurement of your weight and vital signs.
* You will be asked about any side effects you may be having.
* You will be asked about any drugs you may have taken or may be taking.
* Your performance status will be recorded.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for blood sugar tests. If you have a history of diabetes, you will need to fast for 8 hours before these blood sugar tests.

At Weeks 4 and 12:

* You will have a physical exam, including a measurement of your vital signs.
* You will be asked about any side effects you may be having.
* You will be asked about any drugs you may have taken or may be taking.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for blood sugar tests. If you have a history of diabetes, you will need to fast for 8 hours before these blood sugar tests.

At Weeks 8, 16 and then every 2 months after that, and after your last dose of study drugs:

* You will have a physical exam, including a measurement of your vital signs.
* You will be asked about any side effects you may be having.
* You will be asked about any drugs you may have taken or may be taking.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.
* Blood (about 4 teaspoons) will be drawn for biomarker testing (at weeks 8, 16 and 24 only).
* Blood (about 1 teaspoon) will be drawn for blood sugar tests. If you have a history of diabetes, you will need to fast for 8 hours before these blood sugar tests.
* You will have imaging scans to check the status of the disease.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Exemestane is FDA approved and commercially available for the treatment of metastatic breast cancer. Metformin is FDA approved and commercially available for the treatment of diabetes. Everolimus is FDA approved and commercially available to treat metastatic breast cancer, advanced kidney cancer in some patients and a certain type of brain tumor. The use of this drug combination is investigational.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal overweight or obese women with a history of biopsy-proven hormone receptor-positive breast cancer and clinical evidence of metastatic disease. Overweight is defined as body mass index (BMI) of 25 - 29.9 kg/m2 while obese is defined as BMI >/= 30 kg/m2. Postmenopausal status is defined by one of the following: a) no spontaneous menses for over 1 year, in women >/=55 years; b) no spontaneous menses within the past 1 year in women < 55 years with postmenopausal gonadotrophin levels (LH and FSH levels > 40 IU/L) or postmenopausal estradiol levels (by local laboratory range); or c) bilateral oophorectomy.
2. Prior hormonal therapy for metastatic breast cancer is allowed. Patients who develop progressive metastatic disease on a non-steroidal aromatase inhibitor are eligible. Patients who develop metastatic disease while receiving a non-steroidal aromatase inhibitor in the adjuvant setting are eligible.
3. One prior chemotherapy line for metastatic breast cancer is allowed if there is evidence of progressive disease. Patients treated with chemotherapy to best response and no evidence of progression are not eligible.
4. Prior tamoxifen, LH/RH agonist, anastrozole or letrozole therapy in the adjuvant and/or neoadjuvant settings is allowed. Prior adjuvant and/or neoadjuvant chemotherapy is allowed.
5. Patients must have: [1] at least one lesion that can be accurately measured in at least one dimension >/= 20 mm with conventional imaging techniques or >/= 10 mm with spiral CT or MRI; or [2] bone lesions: lytic or mixed (lytic + sclerotic) in the absence of measurable disease; the following will be considered disease progression among these patients: a) the appearance of one or more new lytic lesions in bone; b) the appearance of one or more new lesions outside of bone; c) unequivocal progression of existing bone lesions.
6. Localized radiotherapy, which does not influence the signal of evaluable lesion, is allowed prior to the initiation of study medications.
7. ECOG performance status </= 2.
8. Absolute neutrophil count (ANC) >/= 1000/microliter, platelets >/= 75,000/microliter, hemoglobin >/= 8.5 gm/dL; creatinine clearance >60 mg/dL; bilirubin < 1.5 mg/dL (</= 3 × ULN for patients known to have Gilbert Syndrome); ALT <3 x upper limit of normal (or </= 5 if hepatic metastases are present); alkaline phosphatase < 3 x upper limit of normal; calcium </= 11.0 mg/dL.
9. Fasting serum cholesterol </= 300 mg/dl or 7.75 mmol/L and fasting triglycerides </= 2.5 × ULN. In case one or both of these thresholds are exceeded, the patient can only be included after initiation of statin therapy and when the above mentioned values have been achieved.
10. Bisphosphonate treatment is permitted for the management of bone loss and/or bone metastases.
11. Patients must be competent to give informed consent and to state that they understand the investigational nature of the proposed treatment.

Exclusion Criteria:

1. HER2-overexpressing breast cancer (IHC 3+ staining or in situ hybridization positive).
2. Diabetes mellitus on active treatment or hemoglobin A1C >/= 6.5% or random plasma glucose > 200 mg/dL in patients without known diabetes.
3. Treatment with metformin in the 30 days prior to enrollment.
4. Known hypersensitivity or intolerance to metformin.
5. Previous treatment with exemestane or mTOR inhibitors.
6. Known hypersensitivity to mTOR inhibitors, e.g. sirolimus (rapamycin).
7. History of acromegaly, Cushing's syndrome, Cushing's disease, Addison's disease (treated or untreated).
8. Patients with unstable angina, uncontrolled ischemic cardiac disease or symptomatic congestive heart failure (e.g. Class III or IV New York Heart Association's Functional Classification).
9. Other investigational drugs within the past 3 weeks or concurrently.
10. Patients with known chronic liver diseases (e.g., chronic active hepatitis, and cirrhosis).
11. Another malignancy within 5 years prior to registration, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer.
12. Radiotherapy within four weeks prior to registration except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture which can then be completed within two weeks prior to registration. Patients must have recovered from radiotherapy toxicities.
13. History of brain or other central nervous system metastases.
14. Bilateral diffuse lymphangitic carcinomatosis.
15. Presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement, or any degree of brain or leptomeningeal involvement (past or present), or symptomatic pulmonary lymphangitic spread. Subjects with discrete pulmonary parenchymal metastases are eligible, provided their respiratory function is not compromised as a result of disease.
16. Patients receiving concomitant immunosuppressive agents or chronic corticosteroids use, at the time of study entry except in cases outlined below: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed. Patients on stable low dose of corticosteroids for at least two weeks before enrollment are allowed.
17. Any severe and / or uncontrolled medical conditions such as: Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction </= 6 months prior to enrollment, serious uncontrolled cardiac arrhythmia; Uncontrolled diabetes as defined by fasting serum glucose > 1.5 × ULN; Acute and chronic, active infectious disorders (except for Hep B and Hep C positive patients) and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy; Impairment of gastrointestinal function or who have gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome); Active skin, mucosa, ocular or GI disorders of Grade > 1
18. Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air will be considered to exclude restrictive pulmonary disease, pneumonitis or pulmonary infiltrates.
19. Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A (Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itraconazole, Voriconazole, Ritonavir, Telithromycin) within the last 5 days prior to registration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Valero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from October 2012 to September 2013. The participating subjects must sign the consent document pertaining to the study and meet all the eligibility criteria as mentioned in the protocol, before initiating on the study treatment.
Groups:
- Everolimus + Exemestane + Metformin: Exemestane 25 mg by mouth once a day daily for 28, Everolimus 10 mg by mouth once a day daily for 28, days and Metformin upto 1000 mg by mouth twice a day daily for 28 days cycle.
Period: Overall Study
Arm/Group | Everolimus + Exemestane + Metformin
Started | 23
Completed | 22
Not Completed | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus + Exemestane + Metformin
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 57.2 [37.6 to 70.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The primary end point of this study was progression-free survival (PFS), defined as the time from study enrollment to disease progression or death from any cause, whichever occurred first. Data for PFS were censored at the time of a patient's removal from study. All other analyses were post-hoc and should be regarded as such.
Time Frame: From the registration until disease progression, death, unacceptable toxicity, or withdraw of study consent, whichever occurred first assessed up to 67 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Exemestane + Metformin
Number analyzed (Participants) | 22
months | 6.3 [3.8 to 11.3]

2. Primary Outcome: Compare Progression Free Survival (PFS) Between the Number of Obese and Overweight Participants
Description: The primary end point of this study was progression-free survival (PFS), defined as the time from study enrollment to disease progression or death from any cause, whichever occurred first. Data for PFS were censored at the time of a participants removal from study. Compare PFS between overweight patients (n=11; BMI </=25 kg/m2) and obese patient ( n=11; BMI >/=25 kg/m2) on univariable cox regression analysis.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Compare PFS Between Obese and Overweight Participants: obese patient ( n=11; BMI >/=25 kg/m2) and overweight patients (n=11; BMI </=25 kg/m2)
Arm/Group | Compare PFS Between Obese and Overweight Participants
Number analyzed (Participants) | 22
Participants
  Obese participants | 11
  Overweight participants | 11
Statistical Analysis 1: Comparison: Compare PFS Between Obese and Overweight Participants; Data for PFS were censored at the time of a patient's removal from study. With 40 patients accrued at a rate of 2 patients per month, a one-sided alpha of 5%, and a post- accrual follow up of 3 months, we would have 80% power to detect a median PFS of 12 months as being statistically significantly higher than a historical control median PFS of 7 months. The study terminated early due to lack of efficacy and funds only 22 patients were enrolled in the study; Test type: Non-Inferiority — The study terminated early due to lack of efficacy and funds only 22 patients were enrolled in the study. With 40 patients accrued at a rate of 2 patients per month, a one-sided alpha of 5%, and a post- accrual follow up of 3 months, we would have 80% power to detect a median PFS of 12 months as being statistically significantly higher than a historical control median PFS of 7 months; p = 0.015, Regression, Cox; Cox Proportional Hazard = 0.25, 95% CI 2-sided [0.08 to 0.76]

3. Post Hoc Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from study enrollment to death from any cause. Data on vital status were collected after study completion through May 1, 2018 and were used in the determination of OS.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Exemestane + Metformin
Number analyzed (Participants) | 22
months | 28.8 [17.5 to 59.7]

4. Post Hoc Outcome: Number of Participants With Response
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The clinical benefit rate (CBR) was defined as the proportion of patients with a best overall response of CR, PR or SD (non-CR/non-PD for patients without measurable disease) lasting at least 24 weeks. For patients with a best overall response of CR or PR, the duration of response (DOR) was defined as the time from first documentation of CR or PR to the time of disease progression. Data on the DOR and PFS were censored at the time of a patient's removal from the study. For patients with a best overall response of SD (non-CR/non-PD for patients without measurable disease),the duration of SD (non-CR/non-PD for patients without measurable disease) was defined as the time from study enrollment to the time of disease progression.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus + Exemestane + Metformin
Number analyzed (Participants) | 22
Participants
  Complete Response | 0
  Partial response | 5
  Stable Disease lasting >=24 wks | 7
  Stable Disease lasting <24 wks | 5
  Progressive disease | 5
  Overall response (CR+PR) | 5
  Clinical benefit (CR+PR+SD >/= 24 wks | 12

5. Post Hoc Outcome: Compare Overall Survival (OS) Between the Number of Obese and Overweight Participants
Description: Overall survival (OS) was defined as the time from study enrollment to death from any cause. Data on vital status were collected after study completion through May 1, 2018 and were used in the determination of OS. Compare OS between obese participants ( n=11; BMI >/=25 kg/m2) and overweight participants (n=11; BMI </=25 kg/m2) on univariable cox regression analysis.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Compare OS Between Obese Patient and Overweight Participants: obese patients( n=11; BMI >/=25 kg/m2) and overweight patients (n=11; BMI </=25 kg/m2)
Arm/Group | Compare OS Between Obese Patient and Overweight Participants
Number analyzed (Participants) | 22
Participants
  Obese participants | 11
  Overweight participants | 11
Statistical Analysis 1: Comparison: Compare OS Between Obese Patient and Overweight Participants; Test type: Other; p = 0.31, Regression, Cox; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.22 to 1.62]

ADVERSE EVENTS:
Time Frame: Adverse events collected from the initiation of study drugs until disease progression, death, unacceptable toxicity, or withdraw of study consent, whichever occurred first assessed up to 67 months
Description: There were no deaths. All participants survived.
Arm/Group | Everolimus + Exemestane + Metformin
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Exemestane + Metformin (N=22)
Nausea (Gastrointestinal disorders) | 1
Vomitting (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus + Exemestane + Metformin (N=22)
Nausea (grade 2) (Gastrointestinal disorders) | 3 (3)
Vomitting (grade 2) (Gastrointestinal disorders) | 3 (3)
Diarrhea (grade 2) (Gastrointestinal disorders) | 3 (3)
Fatigue (Investigations) | 6 (6)
Weight loss (Metabolism and nutrition disorders) | 13 (13)
Mucositis (Gastrointestinal disorders) | 10 (10)
AST elevation (Hepatobiliary disorders) | 5 (5)
Hyperglycemia (Endocrine disorders) | 5 (5)
Infection (Infections and infestations) | 4 (4)
ALT elevation (Hepatobiliary disorders) | 3 (3)
Anorexia (General disorders) | 2 (2)
Insomnia(grade 2) (General disorders) | 2 (2)
Rash (grade 2) (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia(grade 2) (Blood and lymphatic system disorders) | 1 (1)
Dyspnea(grade 2) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Fever(grade 2) (General disorders) | 1 (1)
Generalized muscle weakness(grade 2) (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT01627067/Prot_SAP_000.pdf